CLINICAL TRIAL: NCT01954121
Title: An Open-label, Randomized, Parallel-group, Active-controlled Study Comparing the Efficacy and Safety of Levetiracetam to Carbamazepine Used as Monotherapy in Subjects Newly or Recently Diagnosed as Epilepsy and Partial-onset Seizures
Brief Title: Open-label, Randomized, Active-controlled Study of LEV Used as Monotherapy in Patients With Partial-Onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N01364
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Results first posted 2016-08-11 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-07

CONDITIONS: Epilepsy; Partial Seizures
Keywords: Levetiracetam; Keppra; Monotherapy; China; Epilepsy; Partial-onset Seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Levetiracetam; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam (Experimental): Levetiracetam 1000 mg/day
  Interventions: Drug: Levetiracetam
- Carbamazepine (Active Comparator): Carbamazepine 400 mg/day
  Interventions: Drug: Carbamazepine

INTERVENTIONS:
Drug: Levetiracetam — Immediate release film-coated tablets at strengths of 250 mg and 500 mg.
  * Up-titration Period (Week 1 to Week 3): Levetiracetam (LEV) 250 mg twice daily (bid)
  * Stabilization Period and Evaluation Period (Week 3 to Week 30): LEV 500 mg bid
  * Down-titration Period (Week 30 up to Week 33)
  Other Names: Keppra
  Arms: Levetiracetam
Drug: Carbamazepine — Immediate release tablets at a strength of 200 mg.
  * Up-titration Period (Week 1 to Week 3): Carbamazepine- Immediate Release (CBZ-IR) 200 mg once daily (qd)
  * Stabilization Period and Evaluation Period (Week 3 to Week 30): CBZ-IR 200 mg bid
  * Down-titration Period (Week 30 up to Week 33)
  Other Names: Tegretol
  Arms: Carbamazepine

SUMMARY:
To demonstrate the non-inferiority of Levetiracetam (1000 mg/day) versus Carbamazepine Immediate-Release (400 mg/day) used as monotherapy for at least 6 months in a Chinese population with newly or recently diagnosed Epilepsy who are experiencing Partial-Onset Seizures (POS).

ELIGIBILITY:
Inclusion Criteria:

* Subject is of Chinese origin and ≥ 16 years of age
* Subject is newly or recently diagnosed with Epilepsy, having experienced unprovoked Partial-Onset Seizures (POS)
* Subject has experienced at least 2 unprovoked seizures in the year preceding randomization, of which at least 1 unprovoked seizure occurred in the 3 months preceding randomization
* Subject has had an Electroencephalogram (EEG) and a brain Computed Tomography (CT) scan or brain Magnetic Resonance Imaging (MRI) scan consistent with a diagnosis of Epilepsy with POS

Exclusion Criteria:

* Subject tests positive for human leukocyte antigen major histocompatibility complex, class I,B (HLA-B)* 1502 allele
* Subject has a history or presence of seizures of other types than Partial-Onset Seizures (POS)
* Subject has only experienced type IA nonmotor seizures
* Subject has a history or presence of seizures occurring only in clustered patterns
* Subject has a history of clinical or Electroencephalogram (EEG) findings suggestive of Idiopathic Generalized Epilepsy prior to randomization
* Subject has current or previous diagnosis of pseudoseizures, conversion disorders, or other nonepileptic ictal events that could be confused with seizures
* Subject has a history of Status Epilepticus

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (28):
- China (28):
  - 13, Beijing
  - 16, Changchun
  - 10, Chengdu
  - 5, Chengdu
  - 4, Chongqing
  - 11, Guangzhou
  - 1, Guangzhou
  - 20, Guangzhou
  - 26, Guangzhou
  - 24, Hangzhou
  - 22, Harbin
  - 29, Kunming
  - 21, Nanjing
  - 23, Nanjing
  - 6, Nanjing
  - 8, Nanjing
  - 27, Qingdao
  - 14, Shanghai
  - 15, Shanghai
  - 18, Shanghai
  - 2, Shanghai
  - 19, Shijiazhuang
  - 3, Suzhou
  - 9, Taiyuan
  - 25, Tianjin
  - 12, Wuhan
  - 17, Xi'an
  - 7, Xi'an

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in China in September 2013.
Pre-assignment Details: Participant Flow refers to the Randomized Set which consists of all subjects who were randomized in this study.
Groups:
- Levetiracetam: During the Up-Titration period (2 weeks), subjects initiated treatment at half the randomized target dose with Levetiracetam (LEV) 250 mg bid. During Stabilization and Evaluation Period (27 weeks) LEV was taken bid 500 mg.
- Carbamazepine-IR: During the Up-Titration period (2 weeks), subjects initiated treatment at half the randomized target dose with Carbamazepine immediate-release (CBZ-IR) 200 mg qd. During Stabilization and Evaluation (27 weeks) Period CBZ-IR was taken bid 200 mg.
Period: Overall Study
Arm/Group | Levetiracetam | Carbamazepine-IR
Started | 220 | 216
Completed | 93 | 125
Not Completed | 127 | 91
Not completed — Lack of Efficacy | 94 | 41
Not completed — Protocol Violation | 0 | 2
Not completed — Lost to Follow-up | 5 | 6
Not completed — Withdrawal by Subject | 18 | 12
Not completed — Pregnancy | 1 | 1
Not completed — AE, serious fatal | 1 | 0
Not completed — AE, non-serious non-fatal | 5 | 22
Not completed — SAE, non-fatal | 1 | 4
Not completed — Non-compliant with study procedures | 1 | 0
Not completed — Non-compliant patient | 1 | 1
Not completed — Subject did not follow instructions | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics refers to the Safety Set (SS) which consists of all subjects who were randomized and received at least 1 dose of trial medication.
Groups:
- Levetiracetam (Safety Set): During the Up-Titration period (2 weeks), subjects initiated treatment at half the randomized target dose with Levetiracetam (LEV) 250 mg bid. During Stabilization and Evaluation Period (27 weeks) LEV was taken bid 500 mg.
- Carbamazepine-IR (Safety Set): During the Up-Titration period (2 weeks), subjects initiated treatment at half the randomized target dose with Carbamazepine immediate-release (CBZ-IR) 200 mg qd. During Stabilization and Evaluation (27 weeks) Period CBZ-IR was taken bid 200 mg.
Arm/Group | Levetiracetam (Safety Set) | Carbamazepine-IR (Safety Set) | Total Title
Number analyzed (Participants) | 218 | 215 | 433
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 22 | 42
  Between 18 and 65 years | 184 | 186 | 370
  >=65 years | 14 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years]
  mean (standard deviation) | 37.8 (16.2) | 33.3 (14.3) | 35.6 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 94 | 200
  Male | 112 | 121 | 233

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Remaining Seizure Free During the 6-months Evaluation Period
Time Frame: 6-months Evaluation Period (From Week 4 to Week 30)
Population: The Per Protocol Set consisted of all subjects in the Full Analysis Set who entered the Evaluation Period and who did not have any important protocol deviations determined to impact the interpretation of efficacy. Criteria that might impact the assessment of efficacy was determined during a Data Review Meeting before the database lock.
Measure: Number; unit: percentage of subjects
Groups:
- Levetiracetam (Per Protocol Set): During the Up-Titration period (2 weeks), subjects initiated treatment at half the randomized target dose with Levetiracetam (LEV) 250 mg bid. During Stabilization and Evaluation Period (27 weeks) LEV was taken bid 500 mg.
- Carbamazepine-IR (Per Protocol Set): During the Up-Titration period (2 weeks), subjects initiated treatment at half the randomized target dose with Carbamazepine immediate-release (CBZ-IR) 200 mg qd. During Stabilization and Evaluation (27 weeks) Period CBZ-IR was taken bid 200 mg.
Arm/Group | Levetiracetam (Per Protocol Set) | Carbamazepine-IR (Per Protocol Set)
Number analyzed (Participants) | 186 | 171
percentage of subjects | 47.3 | 68.4
Statistical Analysis 1: Comparison: Levetiracetam (Per Protocol Set) vs Carbamazepine-IR (Per Protocol Set); The adjusted absolute difference in treatment group seizure-free proportions (referenced as 'Adjusted difference in proportions' in 'Method of Estimation' below) was derived from the adjusted treatment group proportions of seizure-free subjects. The adjusted proportions were derived from a logistic regression model of seizure freedom using treatment and the categories for the number of seizures in the 3-month period prior to Visit 1 (≤2 seizures and >2 seizures) as covariates; Test type: Non-Inferiority or Equivalence — The non-inferiority margin for the adjusted difference in seizure free proportion in the LEV minus the seizure free proportion in the CBZ-IR group was set to absolute -20% points; adjusted difference in proportions = -22.9, 95% CI 2-sided [-33.1 to -12.6]

2. Secondary Outcome: Proportion of Subjects Retained in the Study for the Duration of the Period Covering the Up Titration Period, Stabilization Period, and Evaluation Period
Time Frame: From Week 1 to Week 30
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Levetiracetam (Per Protocol Set) | Carbamazepine-IR (Per Protocol Set)
Number analyzed (Participants) | 186 | 171
percentage of subjects | 48.4 | 70.2

3. Secondary Outcome: Time to First Seizure or Discontinuation Due to an Adverse Event (AE) / Lack of Efficacy (LOE) During the Evaluation Period
Description: Number of qualifying events is reported because it is the only descriptive measure available from the proportional hazards model, that was applied.
Time Frame: From first day in the Evaluation Period (Week 4) up to end of the Evaluation Period (Week 30)
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Levetiracetam (Per Protocol Set) | Carbamazepine-IR (Per Protocol Set)
Number analyzed (Participants) | 186 | 171
events | 88 | 45

4. Secondary Outcome: Time to First Seizure During the Evaluation Period
Description: as for outcome 3
Time Frame: From first day in the Evaluation Period (Week 4) up to end of the Evaluation Period (Week 30)
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Levetiracetam (Per Protocol Set) | Carbamazepine-IR (Per Protocol Set)
Number analyzed (Participants) | 186 | 171
events | 87 | 39

5. Secondary Outcome: Time to First Seizure During the Period Covering the Up Titration Period, Stabilization Period, and Evaluation Period From the First Dose of Study Drug
Description: as for outcome 3
Time Frame: From Randomization (Week 1) up to Evaluation Visit (Week 30)
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Levetiracetam (Per Protocol Set) | Carbamazepine-IR (Per Protocol Set)
Number analyzed (Participants) | 186 | 171
events | 97 | 57

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from Visit 1 (Week 0) until Safety Follow Up Visit (Week 35).
Description: Adverse Events refer to the Safety Set (SS), which is a subset of the Randomized Set and consisted of all subjects who received at least 1 dose of study medication after randomization, either Levetiracetam or Carbamezepine immediate-release.
Arm/Group | Levetiracetam (Safety Set) | Carbamazepine-IR (Safety Set)
Serious Adverse Events (participants affected / at risk) | 9/218 | 11/215
Other Adverse Events (participants affected / at risk) | 92/218 | 93/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (Safety Set) (N=218) | Carbamazepine-IR (Safety Set) (N=215)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epidural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 2 (2) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (Safety Set) (N=218) | Carbamazepine-IR (Safety Set) (N=215)
Nasopharyngitis (Infections and infestations) | 40 (48) | 32 (42)
Upper respiratory tract infection (Infections and infestations) | 12 (16) | 16 (18)
Urinary tract infection (Infections and infestations) | 11 (12) | 5 (5)
Blood cholesterol increased (Investigations) | 6 (6) | 11 (11)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 11 (11)
White blood cell count decreased (Investigations) | 1 (1) | 11 (14)
Dizziness (Nervous system disorders) | 33 (48) | 18 (29)
Somnolence (Nervous system disorders) | 20 (25) | 7 (8)
Headache (Nervous system disorders) | 19 (33) | 16 (47)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days